CLINICAL TRIAL: NCT05453123
Title: The Effect of Motivational Messages by "WhatsApp" on Adherence to Home Exercise Program Among Middle-aged and Older Adults With Knee Osteoarthritis in Saudi Arabia
Brief Title: The Effect of Motivational Messages by "WhatsApp" on Adherence to Home Exercise Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Lujain Abdullah, physiotherapist, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: kneeOA
Record Dates: First submitted 2022-06-29; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paper-handout arm (Active Comparator): the paper-handout arm is the control group taking the home exercise printed in the paper handout.
  Interventions: Behavioral: telerehabilitation
- intervention arm (Experimental): the intervention arm is the experimental group where they take home exercise and motivational text messages by WhatsUp
  Interventions: Behavioral: telerehabilitation

INTERVENTIONS:
Behavioral: telerehabilitation — examine the effect of the text message platform (WhatsApp) on the adherence to home exercise programs, pain and physical function among middle age and older adults with knee OA in two public hospitals in Riyadh city, Saudi Arabia.

SUMMARY:
This study aims to examine the effect of the text message platform (WhatsApp) on the adherence to home exercise programs, pain and physical function among middle age and older adults with knee OA in two public hospitals in Riyadh city, Saudi Arabia

ELIGIBILITY:
Inclusion Criteria:

Saudi adults aged 45 to 65. Diagnosis of unilateral or bilateral, mild to moderate knee OA

Exclusion Criteria:

Diagnosis of severe knee OA Diagnosis of neurological conditions Diagnosis of cardiopulmonary conditions Diagnosis of mental disorders on wait for surgical intervention.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
Adherence percentage outcome was measured with the self-report | baseline and see the change after 6 weeks
  The participants received an online exercise log via WhatsApp message and were asked to record the date and number of the exercise session

SECONDARY OUTCOMES:
VAS | baseline and see the change after 6 weeks
  a single-item continuous scale composed of a horizontal or vertical line (Hawker et al., 2011). The score is determined by measuring the distance (in mm) on a 10-cm line between the "no pain" (score of 0) anchor and the patient's mark (evaluating their pain), providing a range of scores from 0-to 10. A higher score of 10 indicates higher pain intensity.
WOMAC | baseline and see the change after 6 weeks
  The WOMAC is a disease-specific self-report instrument with 17 items in Physical Function. It has been extensively used; it is valid, reliable, and widely recommended in studies of individuals with knee OA, (score range 0-68 where 68 indicates worse function.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Eickenberg H-U. Letter: Hypoazotemia. Urology. 1975 Aug;6(2):267. doi: 10.1016/0090-4295(75)90734-7. No abstract available. PMID 1145951
- [Background] Al-Arfaj AS, Al-Boukai A. Prevalence of radiographic osteoarthritis of the hands in Saudi Arabia. Rheumatol Int. 2002 Sep;22(5):208-12. doi: 10.1007/s00296-002-0228-5. Epub 2002 Aug 13. PMID 12215868